CLINICAL TRIAL: NCT04751669
Title: Efficacy of Micronutrient Dietary Supplementation in Reducing Hospital Admissions for COVID-19: A Double-blind, Placebo-controlled, Randomized Clinical Trial
Brief Title: Efficacy of a Dietary Supplementation in Reducing Hospital Admissions for COVID-19. Randomized Clinical Trial
Acronym: CoVIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CoVIT Clinical Trial
Record Dates: First submitted 2021-02-11; First posted 2021-02-12 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Covid19
Keywords: Dietary Supplement
MeSH Terms: conditions — COVID-19 | interventions — Vitamins; Trace Elements

STUDY DESIGN:
Intervention Model Description: A double-blind, placebo-controlled, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo tablets with the same external aspect than the dietary supplement, the same administration route, containing only the excipients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micronutrient dietary supplement effervescent tablet (Experimental): Tablet containing:
  * Retinol (Vitamin A) 700 mcg
  * Cholecalciferol (Vitamin D3) 10 mcg
  * Alpha-Tocopherol (Vitamin E) 45 mg
  * Ascorbic acid (vitamin C) 1000 mg
  * Pyridoxine (Vitamin B6) 6.5 mg
  * Cyanocobalamin (Vitamin B12) 9.6 mg
  * Folic acid 400 mg
  * Iron 5 mg
  * Zinc 10 mg
  * Selenium 110 mg
  * Copper 0.9 mg
  * Excipients
  Interventions: Dietary Supplement: Vitamin and trace elements
- Placebo dietary supplement effervescent tablet (Placebo Comparator): Effervescent tablet with only the excipients.
  * Sucralose 13 mg
  * Sodium Chloride 20 mg
  * Potassium Acesulfam 22.5 mg
  * Orange P 55 mg
  * Sodium Carbonate 70 mg
  * Betacarotene 100 mg
  * Malic Acid 800 mg
  * Citric Acid 960 mg
  * Sodium bicarbonate 1,000 mg
  * Isomalt 1,459.50 mg
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin and trace elements — Dietary supplement oral route, once a day, during 14 days
  Arms: Micronutrient dietary supplement effervescent tablet
Dietary Supplement: Placebo — Dietary supplement (placebo) oral route, once a day, during 14 days
  Arms: Placebo dietary supplement effervescent tablet

SUMMARY:
A double-blind, placebo-controlled, randomized clinical trial to assess efficacy of micronutrient dietary supplementation in reducing hospital admissions for COVID-19 and incidence of Long Covid.

We want to assess the need for hospital admission for severe acute respiratory syndrome Corona Virus-2 (SARS-CoV-2) infection in outpatients diagnosed of COVID-19 disease, taking a micronutrient supplementation for 14 days. The outcome Will be measured within 1 month after beginning the study treatment. The patients will be followed-up for a period of 180 days for the incidence of Long Covid

DETAILED DESCRIPTION:
* Type of study/ Design: Randomized, double-blind, placebo-controlled clinical trial.
* Sponsor: Institut d'Investigació en Ciències de la Salut Germans Trias i Pujol / Hospital Universitari Germans Trias i Pujol ( IGTP / HUGTIP)
* Title of the clinical trial: Efficacy of micronutrient dietary supplementation in reducing hospital admissions for COVID-19 and Long Covid: A double-blind, placebo-controlled, randomized clinical trial.
* Protocol code: CoVIT Clinical Trial
* NºClinicaltrials.gov: Pending
* Coordinating researcher: Dra. Teresa-Maria Tomasa-Irriguible.
* Recruiting Center: Germans Trias i Pujol University Hospital (HUGTIP)
* Ethical Committee for clinical Investigation (CEI): Germans Trias i Pujol University Hospital CEI.
* Monitoring: Clinical Research Associate at UPIC (Unitat Polivalent d'Investigació Clínica) Clinical Trial Unit- IGTP
* Study treatments: Dietary supplement with micronutrients and Placebo
* Test phase: Not applicable.
* Main objective: Evaluation of the effectiveness of supplementation with a dietary supplement to improve the need for hospital admission for SARS-CoV-2 infection, and incidence of Long Covid.
* Study pathology: COVID-19.
* Main variable: The need for hospital admission of SARS-CoV-2 documented infection and the incidence of Long Covid
* Study population and total number of patients: Patients of the health system of the Northern Metropolitan Area of Catalan Health Institution with symptoms compatible with SARS-CoV-2 infection. A total of 300 people (150 treated with dietary supplement and 150 with placebo).
* Duration of treatment: 14 days.
* Patients follow-up: 180 days

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent Form signed.
2. Patients with symptoms compatible with COVID-19: cough and fever who not fulfil criteria of hospitalization and will be in outpatient care.
3. Positive polymerase chain reaction (PCR) or transcription-mediated amplification (TMA) test or rapid antigen test for severe acute respiratory syndrome Corona Virus-2 (SARS-CoV-2) or diagnostic test available.
4. Age ≥ 18 years
5. Availability to meet the requirements of the protocol.

Exclusion Criteria:

1. Intake of any micronutrient supplement during the month prior to inclusion.
2. Patients fulfilling hospitalization criteria.
3. Previous allergies to the micronutrient components and excipients.
4. Age ≥ 90 years with any comorbidity (diabetes, hypertension, obesity, heart disease, respiratory disease)
5. Participation in other research that requires experimental intervention (does not include observational studies) in the previous month before signing the informed consent form.
6. Detection by the researcher of lack of knowledge or willingness to participate and comply with all the requirements of the protocol.
7. Any other findings that at the discretion of the researcher may compromise protocol performance or significantly influence the interpretation or results of the effects of the nutritional supplement
8. Pregnancy or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Need for hospital admission | From baseline to 1 month after beginning the study treatment
  The need for hospitalization of documented SARS-CoV-2 infection (positive polymerase chain reaction or transcription-mediated amplification test or antigen test or positive serology or diagnostic test available) over the course of the disease
Incidence of Long Covid. | 6 months after beginning the study treatment
  Incidence of long Covid or symptoms persistence following World Health Organization definition

SECONDARY OUTCOMES:
Micronutrient basal status (Vitamin B1, Vitamin B6, 25-OH-Vitamin D and Folic Acid | Within day 1 at study inclusion
  Evaluation of micronutrient status prior to the nutritional supplement administration (in ng/mL)
Micronutrient basal status (Vitamin B12) | Within day 1 at study inclusion
  Evaluation of micronutrient status prior to the nutritional supplement administration in pg/mL
Micronutrient basal status (Iron, Zinc and Copper ) | Within day 1 at study inclusion
  Evaluation of micronutrient status prior to the nutritional supplement administration in mcg/dL
Micronutrient basal status (Vitamin A and Vitamin E) | Within day 1 at study inclusion
  Evaluation of micronutrient status prior to the nutritional supplement administration in mg/L
Micronutrient basal status (Selenium ) | Within day 1 at study inclusion
  Evaluation of micronutrient status prior to the nutritional supplement administration in mcg/L
Micronutrient basal status (Vitamin C) | Within day 1 at study inclusion
  Evaluation of micronutrient status prior to the nutritional supplement administration in mg/dL
Micronutrient status at hospital admission (Vitamin B1, Vitamin B6, 25-OH-Vitamin D and Folic Acid) | Within the first day of hospital admission
  Evaluation of micronutrient status in patients requiring hospitalization in ng/mL
Micronutrient status at hospital admission ( Vitamin B12) | Within the first day of hospital admission
  Evaluation of micronutrient status in patients requiring hospitalization in pg/mL
Micronutrient status at hospital admission (Iron, Zinc and Copper) | Within the first day of hospital admission
  Evaluation of micronutrient status in patients requiring hospitalization in mcg/dL
Micronutrient status at hospital admission (Vitamin A and Vitamin E) | Within the first day of hospital admission
  Evaluation of micronutrient status in patients requiring hospitalization in mg/L
Micronutrient status at hospital admission (Selenium) | Within the first day of hospital admission
  Evaluation of micronutrient status in patients requiring hospitalization in mcg/L
Micronutrient status at hospital admission (Vitamin C) | Within the first day of hospital admission
  Evaluation of micronutrient status in patients requiring hospitalization in mg/dL
Micronutrient status at end of study (Vitamin B1, Vitamin B6, 25-OH-Vitamin D and Folic Acid) | Within 90 days of the study treatment ending
  Evaluation of micronutrient status after the study treatment in ng/mL
Micronutrient status at end of study (Vitamin B12) | Within 90 days of the study treatment ending
  Evaluation of micronutrient status after the study treatment in pg/mL
Micronutrient status at end of study (Iron, Zinc, and Copper) | Within 90 days of the study treatment ending
  Evaluation of micronutrient status after the study treatment in mcg/dL
Micronutrient status at end of study (Vitamin A and Vitamin E) | Within 90 days of the study treatment ending
  Evaluation of micronutrient status after the study treatment in mg/L
Micronutrient status at end of study (Selenium) | Within 90 days of the study treatment ending
  Evaluation of micronutrient status after the study treatment in mcg/L
Micronutrient status at end of study (Vitamin C) | Within 90 days of the study treatment ending
  Evaluation of micronutrient status after the study treatment in mg/dL
Inflammatory parameters | From baseline to 30 days of the study treatment ending
  Evaluation of C-Reactive Protein, InterLeukin-6 and D-dimer progression during the clinical course of SARS-CoV-2 infection in outpatients
Thromboembolic disease | From baseline to 30 days of the study treatment ending
  Evaluation of thromboembolic disease developed during the clinical course of SARS-CoV-2 infection
Oxygen supplementation | From baseline to the study follow-up period: Maximum 3 months
  Assess the need for oxygen therapy during the clinical course of the infection
High-Flow oxygen supplementation | From baseline to the study follow-up period: Maximum 3 months
  The need for high-flow oxygen therapy during the clinical course of infection
Invasive mechanical ventilation | From baseline to the study follow-up period: Maximum 3 months
  The cumulative incidence of mechanical ventilation requirement for SARS-CoV-2 infection documented
Tracheostomy | From baseline to the study follow-up period: Maximum 3 months
  The need for tracheostomy during the clinical course of SARS-CoV-2 infection
Renal replacement | From baseline to the study follow-up period: Maximum 3 months
  The need for renal replacement therapies during the clinical course of SARS-CoV-2 infection
Death | From baseline to the study follow-up period: Maximum 3 months
  The cumulative incidence of death from SARS-CoV-2 infection is documented
Intensive Care Unit Admission | From baseline to the study follow-up period: Maximum 3 months
  The cumulative incidence of admission to intensive care for SARS-CoV-2 infection documented
Cumulative hospital admission | From baseline to the study follow-up period: Maximum 3 months
  The cumulative incidence of hospital admission for a documented SARS-CoV-2 infection
Hospitalization needs (days) | From baseline to the study follow-up period: Maximum 3 months
  Number of days hospitalized for a SARS-CoV-2 documented infection
Survival | From baseline to the study follow-up period: Maximum 3 months
  Survival
Adverse events | From baseline to the study follow-up period: Maximum 3 months
  Adverse events
Serious Adverse Events | From baseline to the study follow-up period: Maximum 3 months
  Serious adverse events (hospital admissions and mortality)
Persistence (or not) of Covid-19 Clinical Symptoms (directly asking patient for peristence of Neurologic, Psicologic, Digestive, Cardiovascular, Respiratory and Osteomuscular Symptoms). | From baseline to the study follow-up period: Maximum 6 months.
  Assess the Post-Covid19 Persistent Symptoms, directly asking patient for Symptoms at the moment of an On site visit at Day 90 and at thelephonic contact on Day 180.
  Questionnaire to the patient to asess persistent symptoms on the following areas:
  Neurologic: Montreal Cognitive Assessment (Mo-CA-BLIND) and Persistent cefalea Psicologic: Anxiety, depression, sleep and mood transtorns Digestive: dispepsia, diarrea, constipation Cardiovascular: tachicardia, arrhythmia, acute mycardial infarction and Ictus Respiratory: dispnea, chest pain Osteomuscular: astenia, artralgia and myalgia and other symptoms expressed by the patient.
Cognitive status | At baseline and at Day 180.
  Assess the Post-Covid19 cognitive status with MoCA-Blind test.
EQ-5D | At baseline and at Day 180.
  Assess the evolution of quality of life during the study.
  EQ-5D-5L quality of life questionnaire will be administered

CONTACTS AND LOCATIONS:
Overall Officials: Teresa M Tomasa-Irriguible, MD-PhD, Principal Investigator — Hospital Germans Trias i Pujol- Intensive Care Unit
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shakoor H, Feehan J, Al Dhaheri AS, Cheikh Ismail L, Ali HI, Alhebshi SH, Apostolopoulos V, Stojanovska L. Role of vitamin D supplementation in aging patients with COVID-19. Maturitas. 2021 Oct;152:63-65. doi: 10.1016/j.maturitas.2021.03.006. Epub 2021 Mar 16. No abstract available. PMID 33757717